CLINICAL TRIAL: NCT06275009
Title: Effects of Lifestyle and Physical Fitness on Cardiovascular Health: a Cohort Study in Chinese Occupational Population
Brief Title: Chinese Occupational Population Cohort of Lifestyle and Physical Fitness (LiFitChina)
Acronym: LiFitChina
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023-1990
Record Dates: First submitted 2024-02-17; First posted 2024-02-23 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Lifestyle; Physical Fitness; Cardiovascular Diseases
Keywords: Lifestyle; physical fitness; Cardiovascular Diseases; cohort
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence and prevalence of metabolic risk factors such as obesity, hypertension, diabetes, and dyslipidemia, as well as cardiovascular diseases (CVD), are continuously rising among the occupational population in China, primarily comprising the middle-aged and young adults. Unhealthy lifestyles and declining physical fitness are independent risk factors affecting cardiovascular health. Additionally, the level of physical fitness is influenced by postnatal lifestyles. Lifestyle factors related to cardiovascular health in the occupational population encompass various aspects, including smoking, physical activity, diet, sleep, psychological stress, etc. These factors may interact or have a synergistic effect, necessitating a comprehensive assessment.

This project proposes a prospective cohort study design to establish a monitoring cohort for lifestyle and physical fitness among the occupational population. The study will track and follow individuals with or without any CVD metabolic risk factors, collecting information on general status, lifestyle, physical fitness, and health examination data. Exposure factors such as lifestyle and physical fitness will be measured annually, and the occurrence of CVD-related health outcomes will be observed. The aim is to develop a comprehensive evaluation index for cardiovascular health lifestyle, analyze the direct and indirect impacts of lifestyle and physical fitness on the occurrence and development of CVD, and explore potential mediating and moderating effects of physical fitness in the association between lifestyle and cardiovascular health.

ELIGIBILITY:
Inclusion Criteria:

* adults between 18-59 years of age
* occupational staff
* willing to accept long-term follow-up

Exclusion Criteria:

* participants with previous CVD history such as myocardial infarction, stroke and severe aortic stenosis;
* with cancer;
* with congenital genetic diseases, or cannot cooperate with the investigation and follow-up due to acquired diseases, such as congenital heart disease, paralysis, deafness, dementia, mental abnormality, developmental retardation, etc.;
* with exercise contraindications;
* duration of pregnancy;
* refuse to sign the informed consent.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: occupational person free of cardiovascular disease at baseline in China
Sampling Method: Non-Probability Sample
Enrollment: 18512 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2026-12-11 (Estimated); Study Completion 2026-12-11 (Estimated)

PRIMARY OUTCOMES:
the composite end point of new major adverse cardiovascular events | 10 years
  including cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, coronary revascularization and unstable angina pectoris requiring hospitalization

SECONDARY OUTCOMES:
new incidence of each major adverse cardiovascular events | 10 years
  new incidence of cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, coronary revascularization, unstable angina requiring hospitalization and other major adverse cardiovascular events
new incidence of cancer | 10 years
  new incidence of cancer and all-cause death
new incidence of all-cause death | 10 years
  new incidence of all-cause death
level of systolic pressure | 10 years
  The level of systolic pressure measured at each follow-up evaluation time point
level of diastolic pressure | 10 years
  The level of diastolic pressure measured at each follow-up evaluation time point
level of blood lipid | 10 years
  The level of blood lipid measured at each follow-up evaluation time point
level of BMI | 10 years
  The level of BMI (weight and height will be combined to report BMI in kg/m^2) measured at each follow-up evaluation time point
level of maximal oxygen uptake (VO2max) | 10 years
  The level of VO2max which is obtained by submaximal exercise testing on cycle ergometer with two-stage workload to assess cardiorespiratory fitness measured at each follow-up evaluation time point
level of metabolic equivalents (METs) | 10 years
  The level of METs which is obtained by submaximal exercise testing on cycle ergometer with two-stage workload to assess cardiorespiratory fitness measured at each follow-up evaluation time point

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China